CLINICAL TRIAL: NCT07376460
Title: Biological and Proteomic Characterisation of Platelet-rich Plasma (PRP) Before and After Mobilisation of Haematopoietic Stem Cells in Peripheral Blood From Women With Low Ovarian Response (Low Responders) and in Vitro Evaluation in Human Ovarian Cell Models
Brief Title: Proteomic and Biological Characterisation of Plasma for the Study of Changes Following Ovarian Reactivation Treatment
Status: Not yet recruiting | Type: Observational
Sponsor: Instituto Valenciano de Infertilidad, IVI Alicante (Other)
Collaborators: BTI Biotechnology Institute S.L (Unknown); Fundación IVI (Other)
Responsible Party: Sponsor
Other Study IDs: 2510-ALC-124-MM
Record Dates: First submitted 2026-01-22; First posted 2026-01-29 (Actual); Last update posted 2026-02-04 (Actual); Status verified 2026-01

CONDITIONS: Poor Ovarian Response; Ovarian Reactivation
Keywords: Poor ovarian response; ovarian reactivation; StemCell Regenera; ovarian rejuvenation therapy; ovarian failure; Stem cell mobilization; PRP; PRGF; Bone Marrow Derived Stem Cells (BMDSC)

STUDY DESIGN:
Observational Model: Other | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Poor responders undergoing ovarian reactivation StemCell Regenera: Women who present a profile of poor responders meaning they have a poor response towards the ovarian stimulation treatment, yielding a low number of oocytes after oocyte retrieval and moreover want to undergo the ovarian reactivation treatment StemCell Regenera.
  Interventions: Combination Product: Platelet Rich Plasma + BMDSCs mobilization

INTERVENTIONS:
Combination Product: Platelet Rich Plasma + BMDSCs mobilization — This intervention entails, in addition to routine platelet-rich plasma (PRP) isolation, prior mobilization of bone marrow derived stem cells into the peripheral blood using filgrastim, a granulocyte colony-stimulating factor. Consequently, the patient benefits both from the stem cells and their paracrine effects on the ovaries, as well as from the direct effects of intraovarian PRP instillation. Overall, this approach provides multiple benefits derived from two distinct biological sources.

SUMMARY:
The samples used in PRGF treatments owe their effectiveness to the handling, concentration, and preservation of their components, which explains why samples obtained with different platelet-rich plasma preparation systems may vary. At IVIRMA Group, we employ the closed system PRGF-Endoret to process these samples for StemCell Regenera samples obtained after mobilizing stem cells with granulocyte colony-stimulating factor stimulators. According to current regulations, PRP samples are considered medicinal products by AEMPS, requiring knowledge of the composition of processed samples to be administered to the patient. The study and quantification of samples used in StemCell Regenera treatments aim to understand how stem cell mobilization performed through this technique influences the characteristics of PRGF-Endoret. In this context, the present project aims to systematically analyse the proteomic profile of PRP/PRGF before and after haematopoietic stem cell mobilisation in poor-responder patients, and to evaluate its biological impact in vitro using human ovarian cell models. This approach will enable the identification of key factors involved in ovarian activation and regeneration, thereby providing a mechanistic basis for optimising regenerative therapies applied in clinical reproductive medicine. Furthermore, it will contribute scientifically relevant insights to the field of research and to patients themselves.

DETAILED DESCRIPTION:
The study design is based on a comparative analysis of the biological and proteomic profiles of platelet-rich plasma enriched with platelet-derived growth factors (PRP/PRGF) processed using the PRGF Endoret® kit, comparing samples obtained before (PRE) and after (POST) stem cell mobilization. The aim is to define the changes induced by the paracrine effect of bone marrow-derived stem cells (CD34⁺) mobilized into peripheral blood.

ELIGIBILITY:
Inclusion Criteria:

* Patients aged between 18 and 43.
* Patients diagnosed with poor ovarian response (POR) or low ovarian reserve according to Bolonia criteria (ESHRE).
* Patients who are indicated for a StemCell Regenera procedure with the use of granulocyte colony-stimulating factors (Filgrastim).
* Patients who agree to participate and sign the informed consent form.

Exclusion Criteria:

* Patients over the age of 43.
* Patients with only one ovary.
* Patients with an autoimmune or haematological disorder.
* Patients currently undergoing treatment with anticoagulant drugs.
* Patients who are allergic to Filgrastim, the granulocyte colony-stimulating factor.

Ages: 18 Years to 43 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Study Population: Patients from IVI Alicante who decide to undergo the ovarian reactivation treatment "StemCell Regenera" at the clinic for improving ovarian function
Sampling Method: Non-Probability Sample
Enrollment: 10 (Estimated)
Dates: Start 2026-02 (Estimated); Primary Completion 2026-04 (Estimated); Study Completion 2026-06 (Estimated)

PRIMARY OUTCOMES:
Biological and proteomic characterisation of the platelet rich plasma | From enrollment to the end of treatment (4 day treatment) at day 5
  Proteomic and biological characterisation of the platelet rich plasma before and after the peripheral blood mobilization of bone marrow derived stem cells in women with poor ovarian response who undergo the ovarian reactivation treatment StemCell Regenera
In vitro functional studies with human ovarian cells | From enrollment to the end of treatment (4 day treatment) at day 5
  In vitro evaluation of the functional effect of PRP both before and after the stem cell mobilization on peripheral blood over human derived ovarian cells, analysing viability and proliferation parameters

CONTACTS AND LOCATIONS:
Locations (1):
- IVIRMA Alicante, Alicante, Alicante, Spain

REFERENCES:
- [Background] Sfakianoudis K, Simopoulou M, Grigoriadis S, Pantou A, Tsioulou P, Maziotis E, Rapani A, Giannelou P, Nitsos N, Kokkali G, Koutsilieris M, Pantos K. Reactivating Ovarian Function through Autologous Platelet-Rich Plasma Intraovarian Infusion: Pilot Data on Premature Ovarian Insufficiency, Perimenopausal, Menopausal, and Poor Responder Women. J Clin Med. 2020 Jun 10;9(6):1809. doi: 10.3390/jcm9061809. PMID 32532000
- [Background] Zhai J, Yao G, Dong F, Bu Z, Cheng Y, Sato Y, Hu L, Zhang Y, Wang J, Dai S, Li J, Sun J, Hsueh AJ, Kawamura K, Sun Y. In Vitro Activation of Follicles and Fresh Tissue Auto-transplantation in Primary Ovarian Insufficiency Patients. J Clin Endocrinol Metab. 2016 Nov;101(11):4405-4412. doi: 10.1210/jc.2016-1589. Epub 2016 Aug 29. PMID 27571179
- [Background] Zeng X, Du L, Yang H, Wang F. Efficacy and safety of recombinant human granulocyte colony-stimulating factor in patients with poor ovarian response: protocol for a multicentre, randomised, controlled trial. BMJ Open. 2023 Dec 30;13(12):e074135. doi: 10.1136/bmjopen-2023-074135. PMID 38159964
- [Background] Yuan L, Huang W, Bi Y, Chen S, Wang X, Li T, Wei P, Du J, Zhao L, Liu B, Yang Y. G-CSF-mobilized peripheral blood mononuclear cells combined with platelet-rich plasma restored the ovarian function of aged rats. J Reprod Immunol. 2023 Aug;158:103953. doi: 10.1016/j.jri.2023.103953. Epub 2023 May 16. PMID 37209460
- [Background] Tandulwadkar S, Karthick MS. Combined Use of Autologous Bone Marrow-derived Stem Cells and Platelet-rich Plasma for Ovarian Rejuvenation in Poor Responders. J Hum Reprod Sci. 2020 Jul-Sep;13(3):184-190. doi: 10.4103/jhrs.JHRS_130_19. Epub 2020 Oct 27. PMID 33311903
- [Background] Sills ES, Wood SH. Autologous activated platelet-rich plasma injection into adult human ovary tissue: molecular mechanism, analysis, and discussion of reproductive response. Biosci Rep. 2019 Jun 4;39(6):BSR20190805. doi: 10.1042/BSR20190805. Print 2019 Jun 28. PMID 31092698
- [Background] Seckin S, Ramadan H, Mouanness M, Kohansieh M, Merhi Z. Ovarian response to intraovarian platelet-rich plasma (PRP) administration: hypotheses and potential mechanisms of action. J Assist Reprod Genet. 2022 Jan;39(1):37-61. doi: 10.1007/s10815-021-02385-w. Epub 2022 Feb 17. PMID 35175511
- [Background] Santamaria A, Ballester A, Munoz M. Enhancing oocyte activation in women with ovarian failure: clinical outcomes of the Stem Cell Regenera study using G-CSF mobilization of peripheral blood stem cells and intraovarian injection of stem cell factor-enriched platelet rich plasma in real-world-practice. Aging (Albany NY). 2025 Jun 27;17(6):1571-1580. doi: 10.18632/aging.206274. Epub 2025 Jun 27. PMID 40587267
- [Background] Roberts LM, Herlihy N, Reig A, Titus S, Garcia-Milian R, Knight J, Yildirim RM, Margolis CK, Cakiroglu Y, Tiras B, Whitehead CV, Werner MD, Seli E. Transcriptomic landscape of cumulus cells from patients <38 years old with a history of poor ovarian response (POR) treated with platelet-rich plasma (PRP). Aging (Albany NY). 2025 Feb 18;17(2):431-447. doi: 10.18632/aging.206202. Epub 2025 Feb 18. PMID 39976580
- [Background] Reig A, Herraiz S, Pellicer A, Seli E. Emerging follicular activation strategies to treat women with poor ovarian response and primary ovarian insufficiency. Curr Opin Obstet Gynecol. 2021 Jun 1;33(3):241-248. doi: 10.1097/GCO.0000000000000703. PMID 33896920
- [Background] Polonio AM, Garcia-Velasco JA, Herraiz S. Stem Cell Paracrine Signaling for Treatment of Premature Ovarian Insufficiency. Front Endocrinol (Lausanne). 2021 Feb 24;11:626322. doi: 10.3389/fendo.2020.626322. eCollection 2020. PMID 33716956
- [Background] Pellicer N, Cozzolino M, Diaz-Garcia C, Galliano D, Cobo A, Pellicer A, Herraiz S. Ovarian rescue in women with premature ovarian insufficiency: facts and fiction. Reprod Biomed Online. 2023 Mar;46(3):543-565. doi: 10.1016/j.rbmo.2022.12.011. Epub 2022 Dec 20. PMID 36710157
- [Background] Orive G, Anitua E. Platelet-rich therapies as an emerging platform for regenerative medicine. Expert Opin Biol Ther. 2021 Dec;21(12):1603-1608. doi: 10.1080/14712598.2021.1936495. Epub 2021 Jun 7. PMID 34043484
- [Background] Nagy B, Kovacs K, Sulyok E, Varnagy A, Bodis J. Thrombocytes and Platelet-Rich Plasma as Modulators of Reproduction and Fertility. Int J Mol Sci. 2023 Dec 11;24(24):17336. doi: 10.3390/ijms242417336. PMID 38139165
- [Background] Molinaro P, Ballester A, Garcia-Velasco JA, Munoz M, Herraiz S. Impact of bilateral intraovarian platelet-rich plasma in women with poor ovarian response or primary ovarian insufficiency: a retrospective study. Fertil Steril. 2025 Sep;124(3):496-505. doi: 10.1016/j.fertnstert.2025.05.143. Epub 2025 May 14. PMID 40379042
- [Background] Marchesi F, Mengarelli A. Biosimilar Filgrastim in Autologous Peripheral Blood Hematopoietic Stem Cell Mobilization and Post-Transplant Hematologic Recovery. Curr Med Chem. 2016;23(21):2217-29. doi: 10.2174/0929867323666160517115907. PMID 27183986
- [Background] Marchante M, Buigues A, Ramirez-Martin N, Martinez J, Pellicer N, Pellicer A, Herraiz S. Single intraovarian dose of stem cell- and platelet-secreted factors mitigates age-related ovarian infertility in a murine model. Am J Obstet Gynecol. 2023 May;228(5):561.e1-561.e17. doi: 10.1016/j.ajog.2023.01.018. Epub 2023 Jan 24. PMID 36706857
- [Background] Macklon NS, Fauser BC. Aspects of ovarian follicle development throughout life. Horm Res. 1999;52(4):161-70. doi: 10.1159/000023456. PMID 10725781
- [Background] Kyrou D, Kolibianakis EM, Venetis CA, Papanikolaou EG, Bontis J, Tarlatzis BC. How to improve the probability of pregnancy in poor responders undergoing in vitro fertilization: a systematic review and meta-analysis. Fertil Steril. 2009 Mar;91(3):749-66. doi: 10.1016/j.fertnstert.2007.12.077. Epub 2008 Jul 21. PMID 18639875
- [Background] Ivaskiene T, Kaspute G, Bareikiene E, Prentice U. Platelet-Rich Plasma and Electrochemical Biosensors: A Novel Approach to Ovarian Function Evaluation and Diagnostics. Int J Mol Sci. 2025 Mar 5;26(5):2317. doi: 10.3390/ijms26052317. PMID 40076937
- [Background] Hopman RK, DiPersio JF. Advances in stem cell mobilization. Blood Rev. 2014 Jan;28(1):31-40. doi: 10.1016/j.blre.2014.01.001. Epub 2014 Jan 14. PMID 24476957
- [Background] Heyn J, Brauninger S, Becker P, Stoeckmann N, Seidl C, Howe S, Daubert S, Furst D, Schrezenmeier H, Bonig H. Healthy volunteer stem cell donors followed up 10 years after stimulation with biosimilar filgrastim. Transfusion. 2025 Aug;65(8):1418-1426. doi: 10.1111/trf.18317. Epub 2025 Jul 9. PMID 40635295
- [Background] Herraiz S, Romeu M, Buigues A, Martinez S, Diaz-Garcia C, Gomez-Segui I, Martinez J, Pellicer N, Pellicer A. Autologous stem cell ovarian transplantation to increase reproductive potential in patients who are poor responders. Fertil Steril. 2018 Aug;110(3):496-505.e1. doi: 10.1016/j.fertnstert.2018.04.025. Epub 2018 Jun 28. PMID 29960701
- [Background] Herlihy NS, Seli E. The use of intraovarian injection of autologous platelet rich plasma (PRP) in patients with poor ovarian response and premature ovarian insufficiency. Curr Opin Obstet Gynecol. 2022 Jun 1;34(3):133-137. doi: 10.1097/GCO.0000000000000784. PMID 35645011
- [Background] Herlihy NS, Cakiroglu Y, Whitehead C, Reig A, Tiras B, Scott RT Jr, Seli E. Effect of intraovarian platelet-rich plasma injection on IVF outcomes in women with poor ovarian response: the PROVA randomized controlled trial. Hum Reprod. 2024 May 9:deae093. doi: 10.1093/humrep/deae093. Online ahead of print. PMID 38725194
- [Background] Farimani M, Heshmati S, Poorolajal J, Bahmanzadeh M. A report on three live births in women with poor ovarian response following intra-ovarian injection of platelet-rich plasma (PRP). Mol Biol Rep. 2019 Apr;46(2):1611-1616. doi: 10.1007/s11033-019-04609-w. Epub 2019 Feb 5. PMID 30725347
- [Background] Cozzolino M, Herraiz S, Titus S, Roberts L, Romeu M, Peinado I, Scott RT, Pellicer A, Seli E. Transcriptomic landscape of granulosa cells and peripheral blood mononuclear cells in women with PCOS compared to young poor responders and women with normal response. Hum Reprod. 2022 May 30;37(6):1274-1286. doi: 10.1093/humrep/deac069. PMID 35451009
- [Background] Buigues A, Ramirez-Martin N, Martinez J, Pellicer N, Meseguer M, Pellicer A, Herraiz S. Systemic changes induced by autologous stem cell ovarian transplant in plasma proteome of women with impaired ovarian reserves. Aging (Albany NY). 2023 Dec 26;15(24):14553-14573. doi: 10.18632/aging.205400. Epub 2023 Dec 26. PMID 38149997
- [Background] Buigues A, Marchante M, de Miguel-Gomez L, Martinez J, Cervello I, Pellicer A, Herraiz S. Stem cell-secreted factor therapy regenerates the ovarian niche and rescues follicles. Am J Obstet Gynecol. 2021 Jul;225(1):65.e1-65.e14. doi: 10.1016/j.ajog.2021.01.023. Epub 2021 Feb 1. PMID 33539826
- [Background] Buigues A, Diaz-Gimeno P, Sebastian-Leon P, Pellegrini L, Pellicer N, Pellicer A, Herraiz S. Pathways and factors regulated by bone marrow-derived stem cells in human ovarian tissue. Fertil Steril. 2021 Sep;116(3):896-908. doi: 10.1016/j.fertnstert.2021.04.009. Epub 2021 May 8. PMID 33975729
- [Background] Atkinson L, Martin F, Sturmey RG. Intraovarian injection of platelet-rich plasma in assisted reproduction: too much too soon? Hum Reprod. 2021 Jun 18;36(7):1737-1750. doi: 10.1093/humrep/deab106. PMID 33963408
- [Background] Anitua E, Prado R, Azkargorta M, Rodriguez-Suarez E, Iloro I, Casado-Vela J, Elortza F, Orive G. High-throughput proteomic characterization of plasma rich in growth factors (PRGF-Endoret)-derived fibrin clot interactome. J Tissue Eng Regen Med. 2015 Nov;9(11):E1-12. doi: 10.1002/term.1721. Epub 2013 Mar 18. PMID 23505226
- [Background] Barrenetxea G, Celis R, Barrenetxea J, Martinez E, De Las Heras M, Gomez O, Aguirre O. Intraovarian platelet-rich plasma injection and IVF outcomes in patients with poor ovarian response: a double-blind randomized controlled trial. Hum Reprod. 2024 Apr 3;39(4):760-769. doi: 10.1093/humrep/deae038. PMID 38423539